CLINICAL TRIAL: NCT05909527
Title: A Single-arm, Open-label, Single-center Clinical Study: Safety and Efficacy of Anti-CD7 CAR-T in the Treatment of Relapsed or Refractory T Cell Lymphoblastic Acute Leukemia/ Lymphoma
Brief Title: A Clinical Study of CAR-T Treating Relapsed or Refractory T Cell Lymphoblastic Acute Leukemia/ Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-22-004
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: T-Cell Acute Lymphocytic Leukemia
Keywords: T-ALL; CAR T-cell therapy; CD7
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Dose escalation: After enrollment ,Participants complete the PBMC apheresis, then complete the Lymphocyte clearance, and then receive the dose climming test: 0.50E6/kg±20%, 1.00E6/kg±20%、2.00E6/kg±20%.
  Dose Expansion: During or after the dose increase process, if a certain dose group is determined to have preliminary anti-tumor effects and controllable safety, it can be extended at this dose level to further evaluate the tolerance and safety of CD7 CAR-T injection, and to preliminarily evaluate its effectiveness.
  Interventions: Biological: CD7 CAR-T

INTERVENTIONS:
Biological: CD7 CAR-T — A single infusion of autologous CD7 CAR-T cells administered intravenously

SUMMARY:
This study is a single arm, non blind, randomized, single center study aimed at evaluating the safety, pharmacokinetic characteristics, and preliminary efficacy of CD7 CAR-T cell injection in r/r T-ALL/LBL subjects.

DETAILED DESCRIPTION:
This study is a single dose escalation and dose extension study. The main purpose of the IIT clinical trial is to evaluate the safety, tolerance, pharmacokinetic characteristics, and preliminary efficacy of CAR-T cells in r/r T-ALL/LBL subjects. The study includes two parts: the dose increasing stage (Part A) and the dose expanding stage (Part B) of CD7 CAR-T cell injection. The study plans to enroll 30 subjects, of which approximately 12-18 are planned to be enrolled in the dose escalation phase, and the remaining are planned to be enrolled in the dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian understands and voluntarily signs the informed consent form, and is expected to complete the follow-up examination and treatment of the study procedure;
2. Age 2~60 (including threshold), regardless of gender;
3. According to the WHO 2016 standard, the patients with relapsed/refractory acute T-lymphoblastic leukemia/lymphoma (including early pre T-lymphoblastic leukemia) who failed to receive standard treatment or lacked effective treatment methods met any of the following criteria:

1) Recurrence: disease recurrence is confirmed after receiving at least two treatment schemes to achieve complete remission in the past, or disease recurrence occurs after stem cell transplantation to achieve complete remission; 2) Difficult to treat: Have received at least two treatment schemes in the past, and failed to reach CR (for leukemia patients) or PR (for lymphoma patients) after the last treatment, or failed to get remission or develop disease after stem cell transplantation;

4. During screening, the bone marrow examination was definitely diagnosed as CD7 positive by flow cytometry and/or the tumor was definitely diagnosed as CD7 positive by pathological immunohistochemistry, and the positive rate of CD7 was ≥ 70%;

5. The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is less than grade 2 (unless the abnormality is related to the tumor or is judged to be stable by the researcher, which has little impact on the safety or efficacy);

6. The ECOG physical condition score is 0~2 and the expected life span is more than 3 months;

7. With appropriate organ functions:

1. Glutamic alanine transaminase (ALT) and glutamic oxaloacetic transaminase (AST) ≤ 3 times the upper limit of normal value (ULN). The researcher judges that ALT and AST are abnormal due to diseases (such as liver infiltration or bile duct obstruction), and their indicators can be relaxed to ≤ 5 times ULN;
2. Total bilirubin ≤ 1.5 times ULN;
3. Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min;
4. Hemoglobin ≥ 70g/L or maintained at this level after blood transfusion;
5. Indoor oxygen saturation ≥ 92%;
6. Left ventricular ejection fraction (LVEF) ≥ 45%.

Exclusion Criteria:

1. When collecting and preparing CAR-T blood, those with a tumor load greater than 70%;
2. Have malignant tumors other than T-cell hematological malignancies within 5 years, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, breast ductal carcinoma in situ after radical resection cancer.
3. CNS leukemia patients with clinical symptoms.
4. Hepatitis B surface antigen (HBsAg) is positive, hepatitis B core antibody (HBcAb) is positive and the detection of hepatitis B virus (HBV) DNA titer in peripheral blood is not within the normal reference value range; Individuals with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; People who are positive for human immunodeficiency virus (HIV) antibodies; Positive individuals for cytomegalovirus (CMV) DNA testing; Syphilis test positive.
5. Those with a history of severe allergies or known any of the active ingredients, excipients or mouse-derived products contained in the drug, or those allergic to xenogeneic proteins in this trial, including lymphocyte depletion regimens. Severe allergy history is defined as an allergic reaction of grade two or above, and any of the following clinical manifestations occur when an allergic reaction occurs: airway obstruction (runny nose, cough, wheezing, dyspnea), hypercardia tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiration, cardiac arrest.
6. Severe heart disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (refractory Hypertension is defined as: on the basis of improving lifestyle, a reasonable tolerable and sufficient amount of ≥3 kinds of antihypertensive drugs (including diuretics) has been used for > 1 month and the blood pressure has not reached the standard, or the blood pressure can only be achieved effective control after taking ≥4 kinds of antihypertensive drugs.
7. Have unstable systemic disease as judged by the investigator: including but not limited to severe liver, kidney or metabolic disease requiring drug therapy.
8. Those who have received organ transplants or are about to receive organ transplants (except for hematopoietic stem cell transplants).
9. Patients with acute and chronic graft-versus-host disease (GVHD).
10. Patients who received hematopoietic stem cell transplantation within 6 months before screening and who have active GVHD after stopping Immunosuppressive drug therapy.
11. Active autoimmune or inflammatory diseases of the nervous system (eg, Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (eg, cerebral edema) , Posterior Reversible Encephalopathy Syndrome (PRES)).
12. Those who have tumor emergencies (such as spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) before screening or reinfusion and need emergency treatment.
13. The presence of an uncontrolled bacterial, fungal, viral or other infection requiring antibiotic treatment.
14. Those who have undergone major surgical operations (except diagnostic surgery and biopsy) within 4 weeks before clearing the lymph cells, or those who plan to undergo major surgery during the study period, or those whose surgical wounds have not healed completely before enrollment.
15. Those who have received (attenuated) live virus vaccine within 4 weeks before screening.
16. Persons with severe mental illness.
17. Those who are alcoholics or have a history of drug abuse.
18. Pregnant or lactating women, female subjects who plan to become pregnant within 2 years after cell reinfusion, and male subjects whose partners plan to become pregnant within 2 years after cell reinfusion.
19. Patients with contraindications to any research procedure or with other medical conditions that may expose them to unacceptable risks at the discretion of the investigator and/or clinical criteria.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity, DLT | Up to 28 days after CD7 CAR-T infusion
  After the infusion of CD7 CAR-T cells, subjects still experienced adverse events related to or possibly related to CD7 CAR-T cell infusion after optimal supportive treatment
Maximal Tolerable Dose, MTD | Up to 28 days after CD7 CAR-T infusion
  The highest dose for DLT in ≤ 1/6 subjects
Incidence of Treatment-Emergent Adverse Events | Up to 2 years after CD7 CAR-T infusion
  Count the Incidence of adverse events

SECONDARY OUTCOMES:
Complete Response Rate, CRR | Up to 2 years after CD7 CAR-T infusion
  Proportion of subjects who achieved morphological complete response (CR) and complete response with hematologic incomplete recovery (CRi)
Partial Remission Rate, PRR | Up to 2 years after CD7 CAR-T infusion
  Proportion of subjects who achieved a partial response (PR)
Relapse-Free Survival, RFS | Up to 2 years after CD7 CAR-T infusion
  From remission to relapse or death of the subject (including all causes), whether the subject relapsed or died is unknown until the date of the last follow-up examination.
Event Free Survival, EFS | Up to 2 years after CD7 CAR-T infusion
  Counting from the beginning of cell transfusion until treatment failure, recurrence, or death (various causes). Subjects without any of these events were counted up to the last follow-up examination date. For patients without CR or CRi, EFS is calculated from the beginning of cell transfusion until disease progression or death. Based on the initial event.
Concentration of Cytokine after Infusion | Up to 2 years after CD7 CAR-T infusion
  Calculate the change of cytokine level in peripheral blood by flow cytometry after After CD7 CAR-T infusion. Cytokines include IL-2、IL-6、IL-10、IFN-γ.
Concentration of CAR-T cells after Infusion (PK) | Up to 3 months of CAR-T cell infusion, CAR-T cells were not detected for 2 consecutive times.
  CAR-T in peripheral blood after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Junfang Yang, Bachelor, Principal Investigator — Hebei Yanda Hospital
Locations (1):
- Hebei Yanda Hospital, Langfang, Hebei, China